CLINICAL TRIAL: NCT05494333
Title: Correlation Between Pulmonary Functions and Physical Fitness in Children With β-thalassemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Elsayed Abaas Awad, assistant lecture, Cairo University
Other Study IDs: P.T.REC\012\003478
Record Dates: First submitted 2022-07-30; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: β-Thalassemia; Pulmonary Function; Physical Fitness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2: NO INTERVENTION
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — NO intervention

SUMMARY:
The aims of this study are:

1. To determine the correlation between pulmonary functions and physical fitness in children with β-thalassemia.
2. To differentiate between different types of B-thalassemia in both pulmonary functions and physical fitness

DETAILED DESCRIPTION:
Cohort study: cross-sectional design

A) Subjects:

Sample size estimation will be carried out to determine the recruited number of children selected randomly. Each participant's caregiver will sign a consent form authorizing the participation of their children in this study.

They will be selected based on the following:

Inclusion criteria:

* age range from 6 to 12 years
* children with β-thalassemia major and intermediate of both sex and control healthy children of both sex
* They can follow instruction

Exclusive criteria:

Children will be excluded from the study if they have:

* Defined Cardiovascular or respiratory disorders.
* Renal failure
* Visual or hearing impairment, Mentally retarded children
* Myocardial infarction within the last month
* Unstable angina, Recent thoraco-abdominal surgery
* Thoracic or abdominal aneurysm or Current pneumothorax

II) Materials

1. For evaluation of pulmonary functions The measurements that are made include forced expiratory volume in one second (FEV1), forced vital capacity (FVC) and the ratio of the two volumes (FEV1/FVC).
2. For evaluation of physical fitness Aerobic capacity and endurance By 6-Minute Walk Test , 3 minutes step test and Energy expenditure BMI Balance Pediatric balance scale

ELIGIBILITY:
Inclusion Criteria:

* • age range from 6 to 12 years

  * children with β-thalassemia major and intermediate of both sex and control healthy children of both sex
  * They can follow instruction

Exclusion Criteria:

* • Defined Cardiovascular or respiratory disorders.

  * Renal failure
  * Visual or hearing impairment, Mentally retarded children
  * Myocardial infarction within the last month
  * Unstable angina, Recent thoraco-abdominal surgery
  * Thoracic or abdominal aneurysm or Current pneumothorax

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cohort study: cross-sectional design
  A) Subjects:
  Sample size estimation will be carried out to determine the recruited number of children selected randomly. Each participant's caregiver will sign a consent form authorizing the participation of their children in this study
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
assessment of pulmonary functions by spirometer | baseline - one hour for each participant
  measurements difference in vital capacity and minute ventilation
physical fitness | baseline - one hour for each participant
  functional capacity by 6 minute walk test
cardiorespiratory fitness | baseline - one hour for each participant
  measure by 3 minutes step test to monitor recovery of heart rate after stress test

CONTACTS AND LOCATIONS:
Overall Officials: esraa elsayed, Principal Investigator — Cairo University
Locations (1):
- Esraa Elsayed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No